CLINICAL TRIAL: NCT07388251
Title: Comparative Study of the Effect of Intraperitoneal Instillation of Dexmedetomidine Combined With Bupivacaine 0.25% Versus Bupivacaine 0.25% Alone in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Effect of Intraperitoneal Dexmedetomidine Added to Bupivacaine 0.25% Versus Bupivacaine Alone on Postoperative Analgesia in Patients Undergoing Laparoscopic Cholecystectomy
Acronym: DexBupiVsBupi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Kamal Habib, Lecturer of Anesthesia and Intensive Care, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MS 180/ 2025
Record Dates: First submitted 2025-12-17; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Pain Management; Cholelithiasis; Laparoscopic Cholecystectomy
MeSH Terms: conditions — Cholelithiasis | interventions — Bupivacaine; Infusions, Parenteral; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, double-blinded, parallel-group interventional study. Adult patients undergoing elective laparoscopic cholecystectomy are randomly assigned to receive intraperitoneal instillation of a local anesthetic solution with or without an adjuvant. Allocation is concealed using sealed opaque envelopes, and both patients and postoperative assessors are blinded. All participants undergo standardized anesthetic and surgical procedures. Postoperative assessments, including hemodynamic monitoring and pain evaluation using the Visual Analog Scale, are performed at predefined intervals to assess the effects of the intervention. The study evaluates the analgesic efficacy and safety of the tested solutions while maintaining consistent perioperative care.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine 0.25% intraperitoneal instillation (Active Comparator): Patients undergo laparoscopic cholecystectomy and receive intraperitoneal bupivacaine alone. Postoperative pain, hemodynamics, and analgesic requirements are monitored to evaluate standard pain control.
  Interventions: Drug: Bupivacaine 0.25% intraperitoneal
- Bupivacaine 0.25% + Dexmedetomidine 0.5 µg/kg intraperitoneal instillation (Experimental): Patients undergo laparoscopic cholecystectomy and receive intraperitoneal bupivacaine combined with dexmedetomidine. Postoperative pain, hemodynamics, and analgesic requirements are monitored to assess the added analgesic effect of dexmedetomidine.
  Interventions: Drug: Bupivacaine 0.25% + Dexmedetomidine 0.5 µg/kg intraperitoneal

INTERVENTIONS:
Drug: Bupivacaine 0.25% intraperitoneal — Patients receive 20 mL of 0.25% bupivacaine instilled intraperitoneally across the gallbladder bed at the end of laparoscopic cholecystectomy. Standard anesthesia and perioperative care are maintained for all participants.
  Arms: Bupivacaine 0.25% intraperitoneal instillation
Drug: Bupivacaine 0.25% + Dexmedetomidine 0.5 µg/kg intraperitoneal — Patients receive 20 mL of 0.25% bupivacaine combined with 0.5 µg/kg dexmedetomidine instilled intraperitoneally across the gallbladder bed at the end of laparoscopic cholecystectomy. Standard anesthesia and perioperative care are maintained.
  Arms: Bupivacaine 0.25% + Dexmedetomidine 0.5 µg/kg intraperitoneal instillation

SUMMARY:
Laparoscopic cholecystectomy (LC) is the preferred surgical technique for the management of cholelithiasis owing to its advantages over open surgery, including reduced postoperative pain, shorter hospital stay, and faster recovery. Nevertheless, postoperative pain-particularly in the early postoperative period-remains a clinical challenge and may lead to increased analgesic requirements, delayed ambulation, and prolonged hospitalization. Postoperative pain after LC is multifactorial, resulting from peritoneal irritation, pneumoperitoneum-induced diaphragmatic stretching, and residual intraperitoneal carbon dioxide.

Intraperitoneal instillation of local anesthetics has been widely incorporated into multimodal analgesic strategies to reduce postoperative pain and opioid consumption after laparoscopic surgery. Bupivacaine is commonly used for this purpose; however, its limited duration of action has prompted the use of adjuvants to enhance analgesic efficacy. Dexmedetomidine, a selective α2-adrenergic agonist, possesses analgesic, sedative, and opioid-sparing properties with minimal respiratory depression, making it a promising adjunct to local anesthetics.

This randomized, double-blinded clinical trial was conducted at Ain Shams University Hospitals to compare the analgesic efficacy and safety of intraperitoneal dexmedetomidine combined with bupivacaine versus bupivacaine alone in patients undergoing elective laparoscopic cholecystectomy. Thirty adult patients with ASA physical status I-II were randomly allocated into two equal groups. Group A received intraperitoneal bupivacaine 0.25%, while Group B received intraperitoneal bupivacaine 0.25% combined with dexmedetomidine 0.5 µg/kg, instilled over the gallbladder bed at the end of surgery.

The primary outcome was postoperative pain intensity assessed using the Visual Analog Scale (VAS) over the first 24 hours. Secondary outcomes included hemodynamic parameters, oxygen saturation, time to first rescue analgesia, total opioid consumption, and incidence of postoperative adverse events.

The addition of dexmedetomidine to intraperitoneal bupivacaine significantly reduced postoperative pain scores during the early postoperative period, prolonged the time to first rescue analgesia, and markedly decreased opioid consumption without compromising respiratory function. Hemodynamic changes were mild and clinically acceptable, and adverse events were comparable between groups.

In conclusion, intraperitoneal dexmedetomidine combined with bupivacaine provides superior postoperative analgesia and an opioid-sparing effect compared with bupivacaine alone following laparoscopic cholecystectomy, with an acceptable safety profile.

DETAILED DESCRIPTION:
This study was designed as a prospective, randomized, double-blinded clinical trial conducted at Ain Shams University Hospitals, Cairo, Egypt, over a six-month period. The trial aimed to evaluate the perioperative effects of intraperitoneal instillation of local anesthetic solutions with or without an adjuvant in patients undergoing elective laparoscopic cholecystectomy, under standardized anesthetic and surgical conditions. All enrolled patients underwent laparoscopic cholecystectomy performed by the same surgical team using a standardized four-port technique to minimize variability in surgical manipulation and operative time. Pneumoperitoneum was established using carbon dioxide insufflation and maintained at a constant intra-abdominal pressure throughout the procedure. Preoperative preparation included patient education regarding postoperative pain assessment using the 10-point Visual Analog Scale (VAS) one day before surgery. Patients received standardized premedication with oral alprazolam 0.25 mg on the evening before surgery and on the morning of surgery. In the operating room, a peripheral intravenous line was secured using an 18-gauge cannula, and standard monitoring was applied, including five-lead electrocardiography, non-invasive blood pressure measurement, pulse oximetry, and heart rate monitoring. General anesthesia was induced using intravenous fentanyl (2 μg/kg) and propofol until loss of verbal response. Neuromuscular blockade was achieved using atracurium (0.5 mg/kg) to facilitate tracheal intubation. Anesthesia was maintained with sevoflurane in a mixture of oxygen and nitrous oxide, targeting a minimum alveolar concentration of approximately 1.3. Additional doses of atracurium were administered as required, guided by train-of-four monitoring. All patients received standardized intraoperative analgesic and antiemetic prophylaxis. This included intravenous administration of diclofenac 75 mg diluted in 100 mL of normal saline, paracetamol 1 g, ondansetron 4 mg, and dexamethasone 0.1 mg/kg. Local anesthetic infiltration at trocar insertion sites was performed before skin incision. At the completion of the surgical procedure, following gallbladder removal and peritoneal lavage, intraperitoneal instillation of the study solution was performed through the laparoscopic instillation port, with uniform distribution over the gallbladder bed. The study solution was prepared by an anesthesiologist not involved in patient management or postoperative assessment to ensure blinding. The operating surgeon, patients, and investigators responsible for postoperative data collection were unaware of the contents of the instilled solution. At the end of surgery, residual neuromuscular blockade was reversed using neostigmine (0.05 mg/kg) in combination with glycopyrrolate (0.01 mg/kg). Tracheal extubation was performed once standard extubation criteria were met, and patients were transferred to the post-anesthesia care unit (PACU) for routine monitoring. Postoperative management followed a standardized protocol for all patients. Hemodynamic parameters and oxygen saturation were monitored at predefined intervals during the postoperative period. Pain assessment was conducted using the Visual Analog Scale at regular intervals during the first 24 hours following surgery. Rescue analgesia was administered according to a predefined institutional protocol when clinically indicated. Randomization was performed using a computer-generated random sequence, and allocation concealment was ensured through sealed opaque envelopes prepared by an independent investigator. The study maintained double blinding throughout data collection and analysis phases. Data collection was conducted using standardized case report forms. All collected data were anonymized prior to analysis to maintain patient confidentiality. Statistical analysis was performed using the Statistical Package for Social Sciences (SPSS) software, version 23. Continuous variables were summarized using appropriate descriptive statistics, and comparative analyses were conducted using standard parametric or non-parametric tests as applicable. A two-sided p-value of less than 0.05 was considered statistically significant. Ethical approval for the study was obtained from the Ethical Committee of the Faculty of Medicine, Ain Shams University. Written informed consent was obtained from all participants prior to enrollment, in accordance with the Declaration of Helsinki and institutional guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for laparoscopic cholecystectomy.
* ASA I and II.
* Agreement to participate in the study by the participant or his local guardian.

Exclusion Criteria:

* BMI less than 18 or > 30 kg/m2.
* Psychiatric illness.
* Coagulation disorders.
* Those allergic to local anesthetics, or dexmedetomidine.
* Patients with heart block or heart rate less than 50 bpm.
* Intraoperatively, patients who will be converted into open cholecystectomy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-02 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-21 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity measured by Visual Analog Scale (VAS) | From the entry to the PACU up to 24 hours postoperatively
  Pain intensity will be assessed using the 10-point Visual Analog Scale (VAS) at multiple time points: At the entry to the PACU, and at 1, 2, 4, 6, 8, 16, and 24 hours postoperatively. VAS scoring: 0 = no pain, 2-4 = mild pain, 4-6 = moderate pain, 6-8 = severe pain, 8-10 = worst pain imaginable. The mean VAS score during the first 24 postoperative hours will serve as the primary outcome to evaluate analgesic efficacy between study groups.

SECONDARY OUTCOMES:
Mean arterial blood pressure | From the intraperitoneal instillation of local anesthetics and up to 24 hours postoperatively
  Mean arterial blood pressure (MAP), measured in mmHg, Measurements will be obtained immediately after intraperitoneal instillation of local anesthetics, at the end of surgery, on admission to the post-anesthesia care unit (PACU), and at 1, 2, 4, 6, 8, 16, and 24 hours postoperatively.
Heart rate | From the intraperitoneal instillation of local anesthetics and up to 24 hours postoperatively
  Heart Rate (HR), measured in (Beat/minute). Measurements will be obtained immediately after intraperitoneal instillation of local anesthetics, at the end of surgery, on admission to the post-anesthesia care unit (PACU), and at 1, 2, 4, 6, 8, 16, and 24 hours postoperatively.
Peripheral Oxygen Saturation (SpO₂) | From the intraperitoneal instillation of local anesthetics and up to 24 hours postoperatively
  Peripheral Oxygen Saturation (SpO₂), measured in (%). Measurements will be obtained after intraperitoneal instillation of local anesthetics, at the end of surgery, on admission to the post-anesthesia care unit (PACU), and at 1, 2, 4, 6, 8, 16, and 24 hours postoperatively.
Time to first rescue analgesia | From the end of surgery to the administration of the first rescue analgesic.
  The duration in minutes from the end of surgery to the administration of the first rescue analgesic (pethidine 50 mg) will be recorded.
Total pethidine consumption after surgery | Within the first 24 hours postoperatively
  The total amount of pethidine (mg) administered to each patient as rescue analgesia during the first 24 hours postoperatively will be recorded. This outcome evaluates the overall analgesic requirement and opioid-sparing effect of the intraperitoneal interventions.
Adverse events | Within the first 24 hours postoperatively
  Nausea, Vomiting, Pruritis and Pain

CONTACTS AND LOCATIONS:
Overall Officials: Mariam K Habib, MD, Principal Investigator — Ain Shams University
Locations (1):
- intensive care unit Department, Ain Shams University Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) including age, weight, ASA status, FLACC scores, and analgesic consumption will be shared with qualified researchers upon request after publication. Requests will be reviewed by the Principal Investigator, and approved data will be shared via a secure repository. No personal identifiers will be included
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Start Date: Upon publication of the study results. End Date: 5 years after publication.
Access Criteria: Qualified researchers who provide a methodologically sound proposal and have obtained approval from the study investigators will be able to access the de-identified individual participant data and relevant supporting documents. Requests should be submitted via email to the corresponding author, and data will be shared under a data use agreement ensuring confidentiality and proper use.